CLINICAL TRIAL: NCT02435173
Title: An Open-label, Non-randomized, Within-patient Dose-finding Study Followed by a Randomized, Subject, Investigator and Sponsor Blinded Placebo Controlled Study to Assess the Efficacy and Safety of CDZ173 (Leniolisib) in Patients With APDS/PASLI (Activated Phosphoinositide 3-kinase Delta Syndrome/ p110δ-activating Mutation Causing Senescent T Cells, Lymphadenopathy and Immunodeficiency)
Brief Title: Study of Efficacy of CDZ173 in Patients With APDS/PASLI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCDZ173X2201; 2014-003876-22 (EudraCT Number)
Record Dates: First submitted 2015-02-24; First posted 2015-05-06 (Estimated); Results first posted 2022-03-11 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Common Variable Immunodeficiency (CVID), APDS / PASLI
Keywords: APDS; PASLI; PI3Kdelta
MeSH Terms: conditions — Common Variable Immunodeficiency; Activated PI3K-delta Syndrome | interventions — leniolisib

STUDY DESIGN:
Intervention Model Description: Part I of the study was a non-randomized, open-label, within-patient up-titration dose-finding part in 6 participants with APDS/PASLI. Part II was a randomized, subject, investigator and sponsor-blinded, placebo-controlled, fixed dose part investigating 31 participants with APDS/PASLI.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I: CDZ173 (Experimental): Participants consecutively received CDZ173 10 mg twice a day (b.i.d.) from Day 1 to Day 28, CDZ173 30 mg b.i.d. from Day 29 to Day 56 and CDZ173 70 mg b.i.d. from Day 57 to Day 84.
  Interventions: Drug: CDZ173
- Part II: CDZ173 (Experimental): Participants received CDZ173 70 mg b.i.d. from Day 1 to Day 85.
  Interventions: Drug: CDZ173
- Part II: Placebo (Placebo Comparator): Participants received Placebo b.i.d. from Day 1 to Day 85.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CDZ173 — CDZ173 10 and 70 mg capsules for oral administration.
  Other Names: Leniolisib
  Arms: Part I: CDZ173; Part II: CDZ173
Other: Placebo — Placebo capsules for oral administration
  Arms: Part II: Placebo

SUMMARY:
This study was designed to explore CDZ173, a selective PI3Kδ inhibitor, in patients with genetically activated PI3Kδ, i.e., patients with Activated phosphoinositide 3-kinase delta syndrome/ p110δ-activating mutation causing senescent T cells, lymphadenopathy and immunodeficiency (APDS/PASLI).

The study consisted of two parts: Part I was the open label part designed to establish the safety and pharmacokinetics of CDZ173 in the target population, as well as to select the optimal dose to be tested in Part II. Part II was designed to assess efficacy and safety of CDZ173 in the target population.

DETAILED DESCRIPTION:
This was a 2-part (Part I and Part II), Phase 2/3, multi-center study in subjects with APDS/PASLI.

Part I of the study was a non-randomized, open-label, within-patient up-titration dose-finding part in 6 participants with APDS/PASLI. The starting dose was 10 mg followed by 30 mg and 70 mg b.i.d. for 4 weeks at each dose level respectively. Part I consisted of three distinct study periods:

Screening / Baseline visit (Day -50 to Day-1): This period was used to confirm that the study inclusion and exclusion criteria were met. Participants who were deemed eligible for enrollment into the study attended the clinic on Day -1 for baseline assessments prior to randomization.

Treatment period (Day 1 to Day 84): Participants started treatment on Day 1 receiving 10 mg of CDZ173 twice daily (b.i.d.) until Day 28. After a continuous safety review and a review of PK and PD data, participants assessed as satisfactory proceeded to the next dose levels: from Day 29 to Day 56 participants received 30 mg CDZ173 b.i.d. and from Day 57 to Day 84, if assessed as satisfactory, participants received 70 mg CDZ173 b.i.d.

Follow-up (Day 85-114): After completion of the treatment period, participants were followed-up for safety for four weeks until Day 114.

Part II was a randomized, subject, investigator and sponsor-blinded, placebo-controlled, fixed dose part investigating 31 participants with APDS/PASLI. The CDZ173 dose used in this Part was selected based on safety, tolerability, PK and PD data from Part I. Part II consisted of three distinct study periods:

Screening / Baseline visit (Day -50 to Day-1): This period was used to confirm that the study inclusion and exclusion criteria were met. Participants who were deemed eligible for enrollment into the study attended the clinic on Day -1 for baseline assessments prior to randomization.

Treatment period (Day 1 to Day 85): On Day 1, Participants were randomized to one of the two treatment groups in a 2:1 ratio to receive either 70 mg CDZ173 b.i.d. or matching placebo until Day 85.

Follow-up (Day 86-115): On Day 86, a subset of participants rolled over to CCDZ173X2201E1 extension study and were not followed up for safety after end of treatment in CCDZ173X2201. Participants, who did not directly roll over to the extension study, after last treatment dose were followed-up for safety for four weeks until Day 115.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients 12 to 75 years of age (inclusive), who had a documented APDS/PASLI-associated genetic PI3K delta mutation.
* In Part I and Part II, patients must had nodal and/or extranodal lymphoproliferation, and clinical findings and manifestations compatible with APDS/PASLI such as a history of repeated oto-sino-pulmonary infections and/or organ dysfunction (e.g., lung, liver). Additionally, in part II, patients must had at least one measurable nodal lesion on a CT or MRI scan.
* At screening, vital signs (systolic and diastolic blood pressure and pulse rate) were assessed in the sitting position after the patient rested for at least three minutes.

Key Exclusion Criteria:

* Previous or concurrent use of immunosuppressive medication.
* Current use of medication known to be strong inhibitor or moderate or strong inducers of isoenzyme CYP3A, if treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
* Current use of medications that are metabolized by isoenzyme CYP1A2 and have a narrow therapeutic index (drugs whose exposureresponse indicates that increases in their exposure levels by the concomitant use of potent inhibitors may lead to serious safety concerns (e.g., Torsades de Pointes)).
* Administration of live vaccines (this includes any attenuated live vaccines) starting from 6 weeks before study entry, during the study and up to 7 days after the last dose of CDZ173.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study medication and for 2 days after stopping study treatment.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koneti V Rao, MD, Principal Investigator — National Institutes of Health (NIH); Virgil Dalm, MD, Principal Investigator — Erasmus Medical Center; Anna Šedivá, MD, Principal Investigator — Motol University
Locations (10):
- National Institute of Health NIH, Bethesda, Maryland, United States
- Novartis Investigative Site, Minsk, Belarus
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Dresden, Germany
- Novartis Investigative Site, Dublin, Ireland
- Italy (2):
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Brescia
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Upton JEM, Williams KW, Cant A, Santos A, Bana E Costa J, Bradt J, Harrington A, Gwaltney C. Key outcomes in treatment of activated phosphoinositide 3-kinase delta syndrome: An e-Delphi panel study and responder threshold application. PLoS One. 2025 Oct 15;20(10):e0333341. doi: 10.1371/journal.pone.0333341. eCollection 2025. PMID 41091701
- [Derived] Rao VK, Webster S, Sediva A, Plebani A, Schuetz C, Shcherbina A, Conlon N, Coulter T, Dalm VA, Trizzino A, Zharankova Y, Kulm E, Korholz J, Lougaris V, Rodina Y, Radford K, Bradt J, Kucher K, Relan A, Holland SM, Lenardo MJ, Uzel G. A randomized, placebo-controlled phase 3 trial of the PI3Kdelta inhibitor leniolisib for activated PI3Kdelta syndrome. Blood. 2023 Mar 2;141(9):971-983. doi: 10.1182/blood.2022018546. PMID 36399712
- [Derived] Rao VK, Webster S, Dalm VASH, Sediva A, van Hagen PM, Holland S, Rosenzweig SD, Christ AD, Sloth B, Cabanski M, Joshi AD, de Buck S, Doucet J, Guerini D, Kalis C, Pylvaenaeinen I, Soldermann N, Kashyap A, Uzel G, Lenardo MJ, Patel DD, Lucas CL, Burkhart C. Effective "activated PI3Kdelta syndrome"-targeted therapy with the PI3Kdelta inhibitor leniolisib. Blood. 2017 Nov 23;130(21):2307-2316. doi: 10.1182/blood-2017-08-801191. Epub 2017 Sep 29. PMID 28972011
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1058
- See also: A pediatric Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 10 investigative sites in 9 countries.
Pre-assignment Details: The participants were screened within 50 days prior to enrollment. After screening and baseline assessments, the treatment period started on Day 1.
Groups:
- Part I: CDZ173: Participants consecutively received CDZ173 10 mg b.i.d. from Day 1 to Day 28, CDZ173 30 mg b.i.d. from Day 29 to Day 56 and CDZ173 70 mg b.i.d. from Day 57 to Day 84.
- Part II: CDZ173 70 mg: Participants received CDZ173 70 mg b.i.d. from Day 1 to Day 85.
Period: Overall Study
Arm/Group | Part I: CDZ173 | Part II: CDZ173 70 mg | Part II: Placebo
Started (All participants who were enrolled in Part I or randomized in Part II.) | 6 | 21 | 10
Pharmacokinetics (PK) Analysis Set (All enrolled participants with at least one available valid PK concentration measurement, who received CDZ173 study drug and experienced no protocol deviations with relevant impact on PK data.) | 6 | 19 | 0
Pharmacodynamic (PD) Analysis Set (All enrolled participants who received any study drug and with no protocol deviations with relevant impact on PD data.) | 6 | 19 | 8
Completed | 6 | 21 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: CDZ173 | Part II: CDZ173 70 mg | Part II: Placebo | Total
Number analyzed (Participants) | 6 | 21 | 10 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 9 | 5 | 16
  Between 18 and 65 years | 4 | 12 | 5 | 21
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.2 (5.64) | 22.2 (10.00) | 26.7 (13.43) | 23.43 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 6 | 18
  Male | 4 | 11 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 6 | 18 | 7 | 31
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part I: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs, including significant changes from baseline in physical findings, vital signs, electrocardiograms and laboratory values qualifying and reported as AEs. The number of participants in each category (AEs and SAEs) is reported per dose level: CDZ173 10 mg from Day 1 to Day 28, CDZ173 30 mg from day 29 to day 56 and CDZ173 70 mg from day 57 to day 84.
Time Frame: From the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 114 days
Population: All participants enrolled in Part I.
Measure: Count of Participants; unit: Participants
Groups:
- Part I: CDZ173 10 mg: Participants consecutively received CDZ173 10 mg b.i.d. from Day 1 to Day 28, CDZ173 30 mg b.i.d. from Day 29 to Day 56 and CDZ173 70 mg b.i.d. from Day 57 to Day 84.
Arm/Group | Part I: CDZ173 10 mg
Number analyzed (Participants) | 6
Participants
  CDZ173 10 mg AEs | 2
  CDZ173 10 mg SAEs | 0
  CDZ173 30 mg AEs | 2
  CDZ173 30 mg SAEs | 0
  CDZ173 70 mg AEs | 4
  CDZ173 70 mg SAEs | 0

2. Primary Outcome: Part I: CDZ173 Dose Concentration
Description: Venous whole blood samples were collected for the assessment of the dose-PD and the PK/PD relationship of CDZ173 in participants with APDS/PASLI for dose selection in Part II. CDZ173 was determined by a validated Liquid chromatography - Mass spectometry (LC-MS) method; anticipated Lower Limit of Quantification (LLOQ) was 3 ng/mL. Concentrations below the LLOQ were reported as "zero" and no methods for imputation of missing data were used.
Time Frame: Days 1, 29 and 57 (0.25 and 3 h post morning dose) and Day 84
Population: All participants enrolled in Part I
Measure: Mean (Standard Deviation); unit: Nanogram / millilitre
Arm/Group | Part I: CDZ173
Number analyzed (Participants) | 6
Nanogram / millilitre
  Day 1: 0.25 h post-dose | 10.10 (1.10)
  Day 1: 3 h post-dose | 321.00 (115.00)
  Day 29: 0.25 h post-dose | 249.00 (540.00)
  Day 29: 3 h post-dose | 916.00 (185.00)
  Day 57: 0.25 h post-dose | 150.00 (143.00)
  Day 57: 3 h post-dose | 1710.00 (782.00)
  Day 84 | 998.00 (455.00)

3. Primary Outcome: Part I: Percentage of Inhibition of Unstimulated and Stimulated pAkt Levels in B Cells
Description: Phosphorylation of Akt in ex vivo stimulated and unstimulated B cells was quantified at baseline and at the end of the 4-week treatment period for each of the three dose levels. Determination of the percentage (%) of CD20B+ phospho-Akt positive cells after ex vivo stimulation of whole blood was performed by flow cytometry analysis. The percentage of inhibition of pAkt was defined as (-1) * percent change from baseline pAkt value. Unstimulated cells served as controls at each time point. Baseline was defined as the mean of the day -1 value and the pre-dose value on Day 1 when both were available (if one was missing, then baseline was defined as the existing value). A higher percentage of inhibition of stimulated B cells indicates improvement. No methods for imputation of missing data were used.
Time Frame: Baseline, days 29 and 57 (3 and 12 h post-dose) and day 84
Population: All participants who were enrolled in Part I. At each time point, only participants with a derived baseline value and a result at that time point were included.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part I: CDZ173
Number analyzed (Participants) | 6
Percentage
  CD20B Unstimulated: Day 29 - 3 h post-dose | 82.07 (7.25)
  CD20B Stimulated: Day 29 - 3 h post-dose: number analyzed (Participants) | 5
  CD20B Stimulated: Day 29 - 3 h post-dose | 78.00 (7.25)
  CD20B Unstimulated: Day 29 - 12 h post-dose | 50.58 (18.73)
  CD20B Stimulated: Day 29 - 12 h post-dose | 47.14 (7.83)
  CD20B Unstimulated: Day 57 - 3 h post-dose: number analyzed (Participants) | 2
  CD20B Unstimulated: Day 57 - 3 h post-dose | 86.61 (5.26)
  CD20B Stimulated: Day 57 - 3 h post-dose: number analyzed (Participants) | 3
  CD20B Stimulated: Day 57 - 3 h post-dose | 60.98 (54.05)
  CD20B Unstimulated: Day 57 - 12 h post-dose: number analyzed (Participants) | 5
  CD20B Unstimulated: Day 57 - 12 h post-dose | 53.18 (16.59)
  CD20B Stimulated: Day 57 - 12 h post-dose: number analyzed (Participants) | 3
  CD20B Stimulated: Day 57 - 12 h post-dose | 63.65 (21.03)
  CD20B Unstimulated: Day 84: number analyzed (Participants) | 5
  CD20B Unstimulated: Day 84 | 74.35 (11.03)
  CD20B Stimulated: Day 84: number analyzed (Participants) | 4
  CD20B Stimulated: Day 84 | 78.65 (12.00)

4. Primary Outcome: Part II: Change From Baseline in the log10 Transformed Sum of Product of Diameters (SPD) in the Index Lesions
Description: For the assessment of the impact of CDZ173 on lymphadenopathy, participants were scanned in a magnetic resonance imaging (MRI) or a computed tomography (CT) scanner as based on clinical practice and local regulation. MRI or CT imaging of the neck, chest, abdomen and pelvis was performed. Index lesions were selected from measurable nodal and extranodal lesions as per the Cheson methodology. A maximum of six of the largest dominant lesions were selected and documented at baseline and assessed again at the end of treatment. The change in lymph node size was measured using the log10 transformed sum of product of diameters (SPD), the sum of the longest lesion diameter (mm)" and "longest perpendicular diameter (mm)". A lower score indicates index lesions SPD reduction. A negative change from baseline indicates improvement.
Time Frame: Baseline and Day 85
Population: Pharmacodynamic (PD) analysis set, excluding participants with 0 lesion at baseline. Only participants with baseline and end of treatment lymphadenopathy measurements were included.
Measure: Least Squares Mean (Standard Error); unit: Millimeter on Log10 scale
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 18 | 8
Millimeter on Log10 scale | -0.30 (0.04) | -0.06 (0.06)
Statistical Analysis 1: Comparison: Part II: CDZ173 vs Part II: Placebo; Test type: Superiority; p = 0.0012, ANCOVA; Treatment as a fixed effect and log10 transformed baseline SPD as a covariate; Adjusted means difference = -0.24, 95% CI 2-sided [-0.37 to -0.11], Standard Error of Mean 0.06

5. Primary Outcome: Part II: Change From Baseline in Percentage of naïve B Cells Out of Total B Cells
Description: APDS/PASLI patients suffer from dysregulation in B cell function and differentiation with low numbers of naive B cells. Change from baseline in percentage of naïve B cells out of total B cells at the end of treatment was assessed by flow cytometry to evaluate the pharmacodynamic effect of CDZ173 on B cell immunophenotyping. A higher percentage in naïve B out of total B cells is a positive outcome. A positive change from baseline indicates improvement.
Time Frame: Baseline and Day 85
Population: Pharmacodynamic (PD) analysis set. Only participants with a percentage of less than 48% of naive B cells at baseline and with a measured value at Day 85 were included.
Measure: Least Squares Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 8 | 5
Percentage change from baseline | 34.76 (3.08) | -5.37 (3.95)
Statistical Analysis 1: Comparison: Part II: CDZ173 vs Part II: Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Treatment as a fixed effect and baseline as a covariate; Adjusted means difference = 40.13, 95% CI 2-sided [28.51 to 51.75], Standard Error of Mean 5.04

6. Secondary Outcome: Part I & II: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) for CDZ173
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. AUClast was calculated from plasma concentration-time data using non-compartmental methods. AUClast was calculated at the first day of every CDZ173 dose level (10, 30 and 70 mg) for Part I and (70 mg) for Part II. No methods for imputation of missing data were used.
Time Frame: Part I: Days 1, 29 and 57 / Part II: Day 1
Population: Pharmacokinetics (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: Hour * nanogram / millilitre
Arm/Group | Part I: CDZ173 | Part II: CDZ173
Number analyzed (Participants) | 6 | 19
Hour * nanogram / millilitre
  Day 1 | 1760.0 (441.0) | 10400.0 (2800.0)
  Day 29: number analyzed (Participants) | 6 | 0
  Day 29 | 4760.0 (816.0) |
  Day 57: number analyzed (Participants) | 6 | 0
  Day 57 | 10800.0 (3310.0) |

7. Secondary Outcome: Part I & II: Maximum Observed Plasma Concentration (Cmax) for CDZ173
Description: Venous whole blood samples were collected for activity-based pharmacokinetics characterization. Cmax was calculated from plasma concentration-time data using non-compartmental methods. Cmax was calculated at the first day of every CDZ173 dose level (10, 30 and 70 mg) for Part I and (70 mg) for Part II. No methods for imputation of missing data were used.
Time Frame: Part I: Days 1, 29 and 57 / Part II: Day 1
Population: Pharmacokinetics (PK) Analysis Set
Measure: Mean (Standard Deviation); unit: Nanogram / millilitre
Arm/Group | Part I: CDZ173 | Part II: CDZ173
Number analyzed (Participants) | 6 | 19
Nanogram / millilitre
  Day 1 | 393.0 (137.0) | 2150.0 (576.0)
  Day 29: number analyzed (Participants) | 6 | 0
  Day 29 | 1060.0 (222.0) |
  Day 57: number analyzed (Participants) | 6 | 0
  Day 57 | 2540.0 (747.0) |

8. Secondary Outcome: Part I & II: Mental Component Summary (MCS) and Physical Component Summary (PCS) From Short Form 36 (SF-36) Survey
Description: The SF-36 is a widely used and extensively studied instrument to measure health-related quality of life (HRQoL) among healthy subjects and patients with acute and chronic conditions. It consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The subscales are aggregated to derive two overall summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS) scores. PCS and MCS scores range from 0 to 100 with a higher score indicating a more favorable health state (range = 0 "worst" - 100 "best"). No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 29, 57 and 84 / Part II: Baseline and Days 29, 57 and 85
Population: Pharmacodynamic (PD) analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 6 | 19 | 8
Score on a scale
  Day -1: Mental Component Summary | 47.94 (8.22) | 47.36 (7.98) | 45.94 (8.14)
  Day -1: Physical Component Summary | 47.54 (9.24) | 44.49 (7.08) | 44.06 (8.59)
  Day 29: Mental Component Summary | 47.94 (8.22) | 49.98 (8.06) | 49.52 (6.70)
  Day 29: Physical Component Summary | 47.54 (9.24) | 47.87 (7.66) | 44.62 (7.57)
  Day 57: Mental Component Summary | 47.94 (8.22) | 49.12 (8.17) | 45.92 (7.31)
  Day 57: Physical Component Summary | 47.54 (9.24) | 47.04 (7.30) | 47.20 (9.75)
  Day 84 (Part I) / Day 85 (Part II): Mental Component Summary | 47.94 (8.22) | 49.22 (8.17) | 47.32 (8.73)
  Day 84 (Part I) / Day 85 (Part II): Physical Component Summary | 47.54 (9.24) | 47.59 (6.22) | 47.48 (8.48)

9. Secondary Outcome: Part I & II: Overall Work Impairment Due to Health Score From Work Productivity Activity Impairment and Classroom Impairment Questionnaire (WPAI-CIQ)
Description: The Work Productivity Activity Impairment (WPAI) questionnaire measures the amount of absence or presence for work attendance and daily work activity impairment attributable to APDS/PASLI. As younger participants (age 12 and above) were enrolled in the study the WPAI-CIQ was used for all participants as it also measures the amount of absence or presence for school attendance and daily classroom activity impairment. Participants responded for classroom or work-related questions depending on their situation. WPAI-CIQ consists of 10 questions that yield 4 types of scores: absenteeism, presenteeism, work/classroom productivity loss and activity impairment. The Overall work impairment due to health (%) score ranges from 0 to 100% with 100% indicating total work impairment and 0% no impairment at all. No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 29, 57 and 84 / Part II: Baseline and Days 29, 57 and 85
Population: Pharmacodynamic (PD) analysis set. Only the participants that responded the work-related questions from the WPAI-CIQ and with a value at both baseline and that time point were included.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 2 | 9 | 2
Percentage
  Baseline | 25.00 (35.36) | 51.25 (37.23) | 5.00 (7.07)
  Day 29: number analyzed (Participants) | 1 | 9 | 2
  Day 29 | 44.00 (0) | 35.31 (23.12) | 5.00 (7.07)
  Day 57: number analyzed (Participants) | 1 | 8 | 2
  Day 57 | 62.31 (0) | 35.49 (24.70) | 10.00 (14.14)
  Day 84 (Part I) / Day 85 (Part II) | 44.41 (7.90) | 35.59 (31.85) | 25.00 (7.07)

10. Secondary Outcome: Part I & II: Overall Classroom Impairment Due to Health Score From the Work Productivity Activity Impairment and Classroom Impairment Questionnaire (WPAI-CIQ)
Description: The Work Productivity Activity Impairment (WPAI) questionnaire measures the amount of absence or presence for work attendance and daily work activity impairment attributable to APDS/PASLI. As younger participants (age 12 and above) were enrolled in the study the WPAI-CIQ was used for all participants as it also measures the amount of absence or presence for school attendance and daily classroom activity impairment. Participants responded for classroom or work-related questions depending on their situation. WPAI-CIQ consists of 10 questions that yield 4 types of scores: absenteeism, presenteeism, work/classroom productivity loss and activity impairment. The Overall classroom impairment due to health (%) score ranges from 0 to 100% with 100% indicating total classroom impairment and 0% no impairment at all. A higher percentage indicates a negative outcome. No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 29, 57 and 84 / Part II: Baseline and Days 29, 57 and 85
Population: Pharmacodynamic (PD) analysis set. Only the participants that responded the classroom-related questions from the WPAI-CIQ and with a value at both baseline and that time point were included.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 3 | 5 | 4
Percentage
  Baseline | 65.68 (33.49) | 47.33 (44.75) | 23.75 (30.92)
  Day 29: number analyzed (Participants) | 3 | 2 | 4
  Day 29 | 57.30 (18.09) | 0.00 (0) | 22.65 (24.37)
  Day 57: number analyzed (Participants) | 2 | 2 | 4
  Day 57 | 70.13 (18.68) | 12.14 (3.03) | 22.40 (26.16)
  Day 84 (Part I) / Day 85 (Part II): number analyzed (Participants) | 3 | 1 | 2
  Day 84 (Part I) / Day 85 (Part II) | 68.52 (18.74) | 51.00 (0.00) | 5.00 (7.07)

11. Secondary Outcome: Part I & II: Physician's Global Assessment (PGA)
Description: In the physician's global assessment questionnaire the Investigator rated the disease activity of their patient using 100 mm Visual analogue Scale (VAS) ranging from "no disease activity" (0) to "maximal disease activity" (100). To enhance objectivity, the physician was not aware of the specific patient's global assessment, when performing his own assessment on that patient. No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 29, 57 and 84 / Part II: Baseline and Days 29, 57 and 85
Population: Pharmacodynamic (PD) analysis set. At each time point, only participants with a value at both baseline and that time point were included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 6 | 19 | 8
Score on a scale
  Baseline | 34.7 (17.07) | 47.10 (17.65) | 41.38 (17.78)
  Day 29: number analyzed (Participants) | 6 | 18 | 8
  Day 29 | 21.8 (9.70) | 38.81 (23.73) | 29.75 (9.99)
  Day 57 | 22.5 (13.55) | 34.02 (18.89) | 24.13 (18.34)
  Day 84 (Part I) / Day 85 (Part II) | 8.8 (4.12) | 26.70 (22.82) | 25.88 (16.15)

12. Secondary Outcome: Part I & II: Patient's Global Assessment (PtGA)
Description: In the patient's global assessment questionnaire patients are asked about their APDS/PASLI related well-being using 100 mm visual analogue scale (VAS) ranging from "very poor" (0) to "very good" (100). No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 29, 57 and 84 / Part II: Baseline and Days 29, 57 and 85
Population: Pharmacodynamic (PD) analysis set
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 6 | 19 | 8
Score on a Scale
  Baseline | 62.0 (21.90) | 54.53 (21.47) | 62.50 (26.56)
  Day 29 | 65.0 (22.21) | 68.37 (19.31) | 57.75 (24.03)
  Day 57 | 67.5 (21.83) | 64.79 (19.61) | 69.50 (21.93)
  Day 84 (Part I) / Day 85 (Part II) | 72.5 (13.37) | 67.58 (16.57) | 60.25 (23.66)

13. Secondary Outcome: Part I & II: High Sensivity C Reactive Protein (hsCRP) as Biomarker for Systemic Inflammation
Description: High Sensitivity C reactive protein is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. HsCRP was measured in serum using a latex immunochemilunminometric assay (ICMA). No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 1, 15, 29, 57, 84 / Part II: Baseline and Days 1, 15, 29, 57, 85
Population: Pharmacodynamic (PD) analysis set. At each time point, only participants with a value at that time point were included (no imputation for missing data).
Measure: Mean (Standard Deviation); unit: Milligram / liter
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 6 | 19 | 8
Milligram / liter
  Baseline: number analyzed (Participants) | 6 | 4 | 2
  Baseline | 2.49 (1.29) | 10.58 (17.84) | 5.70 (2.19)
  Day 1: number analyzed (Participants) | 6 | 4 | 2
  Day 1 | 2.43 (1.43) | 8.95 (14.56) | 7.85 (4.88)
  Day 15: number analyzed (Participants) | 6 | 18 | 7
  Day 15 | 0.93 (0.70) | 9.19 (23.12) | 2.06 (1.02)
  Day 29: number analyzed (Participants) | 6 | 18 | 8
  Day 29 | 0.77 (0.36) | 5.55 (11.21) | 2.40 (1.75)
  Day 57: number analyzed (Participants) | 6 | 18 | 8
  Day 57 | 1.20 (0.71) | 6.57 (9.18) | 8.90 (16.66)
  Day 84 (Part I) / Day 85 (Part II): number analyzed (Participants) | 5 | 18 | 8
  Day 84 (Part I) / Day 85 (Part II) | 2.82 (4.11) | 7.54 (18.37) | 2.65 (1.79)

14. Secondary Outcome: Part I & II: Lactate Dehydrogenase (LDH) as Biomarker for Systemic Inflammation
Description: Lactate dehydrogenase is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. LDH was measured in serum using a latex immunochemilunminometric assay (ICMA). No methods for imputation of missing data were used.
Time Frame: Part I: Baseline and Days 1, 15, 29, 57, 84 / Part II: Baseline and Days 1, 15, 29, 57, 85
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units / liter
Arm/Group | Part I: CDZ173 | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 6 | 19 | 8
Units / liter
  Baseline | 130.42 (18.28) | 172.92 (72.25) | 169.38 (41.95)
  Day 1: number analyzed (Participants) | 6 | 17 | 7
  Day 1 | 132.17 (23.10) | 170.88 (72.28) | 175.71 (53.72)
  Day 15: number analyzed (Participants) | 6 | 18 | 7
  Day 15 | 132.17 (11.44) | 190.94 (71.54) | 155.14 (48.09)
  Day 29: number analyzed (Participants) | 6 | 18 | 8
  Day 29 | 125.17 (9.85) | 227.17 (163.41) | 185.25 (51.62)
  Day 57: number analyzed (Participants) | 6 | 19 | 7
  Day 57 | 135.50 (17.66) | 193.11 (64.75) | 167.14 (40.45)
  Day 84 (Part I) / Day 85 (Part II): number analyzed (Participants) | 5 | 19 | 8
  Day 84 (Part I) / Day 85 (Part II) | 142.60 (18.53) | 190.63 (57.62) | 179.13 (73.96)

15. Secondary Outcome: Part II: Beta2 Microglobulin as Biomarker for Systemic Inflammation
Description: Beta2 microglobulin is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. Beta2 microglobulin was measured in serum using a latex immunochemilunminometric assay (ICMA). No methods for imputation of missing data were used.
Time Frame: Baseline and Days 1, 15, 29, 57, 85
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milligram / liter
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Milligram / liter
  Baseline | 2.46 (0.87) | 2.32 (0.96)
  Day 1 | 2.43 (0.88) | 2.31 (0.95)
  Day 15: number analyzed (Participants) | 18 | 7
  Day 15 | 2.10 (1.03) | 2.31 (1.09)
  Day 29: number analyzed (Participants) | 18 | 8
  Day 29 | 2.02 (1.17) | 3.21 (1.61)
  Day 57 | 1.90 (0.72) | 2.42 (1.17)
  Day 85 | 2.01 (1.04) | 2.57 (1.19)

16. Secondary Outcome: Part II: Ferritin as Biomarker for Systemic Inflammation
Description: Ferritin is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. Ferritin was measured in serum using a Electrochemiluminescence immunoassay (ECLIA). No methods for imputation of missing data were used.
Time Frame: Baseline and Days 1, 15, 29, 57, 85
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Microgram / liter
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Microgram / liter
  Baseline: number analyzed (Participants) | 18 | 8
  Baseline | 139.16 (399.73) | 62.05 (81.65)
  Day 1: number analyzed (Participants) | 18 | 8
  Day 1 | 142.67 (411.57) | 61.34 (82.04)
  Day 15: number analyzed (Participants) | 17 | 7
  Day 15 | 146.99 (494.88) | 24.61 (17.41)
  Day 29: number analyzed (Participants) | 16 | 8
  Day 29 | 187.65 (641.16) | 48.43 (61.83)
  Day 57: number analyzed (Participants) | 18 | 8
  Day 57 | 199.97 (657.31) | 51.40 (64.95)
  Day 85: number analyzed (Participants) | 18 | 8
  Day 85 | 139.42 (368.68) | 63.16 (56.64)

17. Secondary Outcome: Part II: Fibrinogen as Biomarker for Systemic Inflammation
Description: Fibrinogen is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. Fibrinogen was measured in serum using an Electrochemiluminescence immunoassay (ECLIA). No methods for imputation of missing data were used.
Time Frame: Baseline and Days 1, 15, 29, 57, 85
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Gram / liter
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Gram / liter
  Baseline | 2.66 (0.76) | 2.68 (0.44)
  Day 1 | 2.61 (0.81) | 2.65 (0.42)
  Day 15: number analyzed (Participants) | 17 | 7
  Day 15 | 2.65 (0.62) | 2.67 (0.42)
  Day 29: number analyzed (Participants) | 18 | 8
  Day 29 | 2.53 (0.54) | 2.66 (0.58)
  Day 57 | 3.01 (0.68) | 2.83 (1.13)
  Day 85 | 2.81 (0.57) | 2.61 (0.57)

18. Secondary Outcome: Part II: Erythrocyte Sedimentation Rate (ESR) as Biomarker for Systemic Inflammation
Description: Erythrocyte sedimentation rate (ESR) is a blood test biomarker for inflammation in the body. Sequential blood samples were collected in all participants. ESR was measured in whole blood using the Westergren method. No methods for imputation of missing data were used.
Time Frame: Baseline and Days 1, 15, 29, 57, 85
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimeter / hour
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Millimeter / hour
  Baseline: number analyzed (Participants) | 16 | 8
  Baseline | 28.09 (19.79) | 25.44 (24.88)
  Day 1: number analyzed (Participants) | 16 | 8
  Day 1 | 26.88 (19.33) | 25.13 (24.51)
  Day 15: number analyzed (Participants) | 14 | 7
  Day 15 | 19.50 (13.52) | 16.00 (12.21)
  Day 29: number analyzed (Participants) | 15 | 8
  Day 29 | 18.33 (13.80) | 26.00 (25.26)
  Day 57: number analyzed (Participants) | 17 | 8
  Day 57 | 18.06 (15.36) | 27.88 (23.04)
  Day 85: number analyzed (Participants) | 17 | 8
  Day 85 | 16.35 (15.99) | 19.63 (18.03)

19. Secondary Outcome: Part II: 3D Volume of Index Lesions
Description: Participants were scanned in a magnetic resonance imaging (MRI) or a computed tomography (CT) scanner as based on clinical practice and local regulation. MRI or CT imaging of the neck, chest, abdomen and pelvis was performed. The 3D volume of index lesions was identified as per the Cheson criteria. A reduction of the 3D volume of the index lesions indicated a positive outcome.
Time Frame: Baseline and Day 85
Population: Pharmacodynamic (PD) analysis set.
Measure: Mean (Standard Deviation); unit: Millimeter^3
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Millimeter^3
  Baseline | 20142.12 (15617.13) | 37123.69 (67325.94)
  Day 85 | 7858.08 (6290.98) | 40169.28 (81844.45)

20. Secondary Outcome: Part II: 3D Volume of the Spleen
Description: Participants were scanned in a magnetic resonance imaging (MRI) or a computed tomography (CT) scanner as based on clinical practice and local regulation. MRI or CT imaging of the spleen was performed and its 3D volume was identified as per the Cheson criteria. A reduction of the spleen volume indicated a positive outcome.
Time Frame: Baseline and Day 85
Population: Pharmacodynamic (PD) analysis set.
Measure: Mean (Standard Deviation); unit: Millimeter^3
Arm/Group | Part II: CDZ173 | Part II: Placebo
Number analyzed (Participants) | 19 | 8
Millimeter^3
  Baseline | 586448.74 (311482.61) | 448456.15 (328641.78)
  Day 85 | 411130.98 (193977.46) | 480333.09 (445371.99)

ADVERSE EVENTS:
Time Frame: Part I and Part II: Adverse events (AEs) were reported from the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 114 days for Part I and 115 days for Part II. For the subset of participants in Part II that rolled over to the extension study (CCDZ173X2201E1) directly after the last treatment dose in Part II, AEs were reported from the start of treatment to end of treatment, assessed up to maximum duration of 85 days.
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment. For Part I AEs were reported based on the CDZ173 dose level received when AE started. Therefore, the 30 days post treatment were only applicable for the CDZ173 70 mg arm.
Groups:
- Part I: CDZ173 10 mg: Participants received CDZ173 10 mg b.i.d. from Day 1 to Day 28.
- Part I: CDZ173 30 mg: Participants received CDZ173 30 mg b.i.d. from Day 29 to Day 56.
- Part I: CDZ173 70 mg: Participants received CDZ173 70 mg b.i.d. from Day 57 to Day 84.
- Part I: Total: Participants consecutively received CDZ173 10 mg b.i.d. from Day 1 to Day 28, CDZ173 30 mg b.i.d. from Day 29 to Day 56 and CDZ173 70 mg b.i.d. from Day 57 to Day 84.
Arm/Group | Part I: CDZ173 10 mg | Part I: CDZ173 30 mg | Part I: CDZ173 70 mg | Part I: Total | Part II: CDZ173 70 mg | Part II: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 3/21 | 2/10
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 4/6 | 4/6 | 18/21 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: CDZ173 10 mg (N=6) | Part I: CDZ173 30 mg (N=6) | Part I: CDZ173 70 mg (N=6) | Part I: Total (N=6) | Part II: CDZ173 70 mg (N=21) | Part II: Placebo (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dependence on oxygen therapy (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: CDZ173 10 mg (N=6) | Part I: CDZ173 30 mg (N=6) | Part I: CDZ173 70 mg (N=6) | Part I: Total (N=6) | Part II: CDZ173 70 mg (N=21) | Part II: Placebo (N=10)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Methylenetetrahydrofolate reductase gene mutation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Episcleritis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vascular device occlusion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Groin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 5 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT02435173/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT02435173/SAP_001.pdf